CLINICAL TRIAL: NCT03107585
Title: Bilateral Intermediate Cervical Plexus Block Under Ultrasound for Thyroid Surgery: Impact on Perioperative Opioid Consumption
Brief Title: Intermediate Cervical Block Under Ultrasound for Thyroid Surgery: Impact on Per and Postoperative Opioid Consumption
Acronym: ICPBUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Mahdia (Other)
Responsible Party: Principal Investigator, Majdoub Ali MD, Clinical Professor, University Hospital, Mahdia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBTCpood
Record Dates: First submitted 2016-01-13; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Local Anesthesia; Analgesia Disorder
Keywords: cervical plexus block; thyroidectomy; opioid consumption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bilateral cervical plexus block (GP1) (Experimental): arm intervention GP1 : after skin disinfection and oral premedication , ultrasound guided cervical bilateral bloc ,with10 ml of bupivacaine 0.25 was realized in each side of deep cervical space; then general anesthesia was performed with local protocol
  Interventions: Procedure: bilateral cervical plexus block
- control(GP2) (Placebo Comparator): GP2 control no specific intervention only general anesthesia was performed with local protocol
  Interventions: Procedure: bilateral cervical plexus block

INTERVENTIONS:
Procedure: bilateral cervical plexus block — with a linear probe and after disinfection vascular neck axis are identified at first. At the cricoid cartilage we conducted an apical scan to locate the carotid bifurcation.at this level is carried out a lateral translation to the visibility of the deep cervical space below the sternocleidomastoidien muscle then a needle 50 is introduced in plane. we proceed in inundation of cervical space
  Other Names: GP1

SUMMARY:
The investigators included prospectively 35 patients undergoing an intermediate cervical block under ultrasound (GP1) before a thyroidectomy ,compared to a group of 35 patients without a block (GP2).

DETAILED DESCRIPTION:
The investigators performed prospective trial with 70 patients randomized in two groups each of 35:

* Group 1 (GP1): bilateral echo-guided intermediate cervical plexus bloc (ICB) by 10 ml of isobaric Bupivacaine (0.25%).
* Group 2 (GP2): control.

Ten minutes after ICB, general anesthesia was realised. Total dose of Remifentanil is calculated upon awakening, the postoperative pain is determined by visual analog scale from 0 to 10 (VAS) statements to H0, H2, H4, H6, H12 and H24. Whenever VAS is greater than or equal to 4, a morphine titration was administered.

Total dose consumption, side effects and satisfaction are noted at the end of protocol.

ELIGIBILITY:
Inclusion Criteria:

* candidate for thyroidectomy
* reoperation l

Exclusion Criteria:

* no consent
* BMI> 34
* allergy to any of the products used
* reoperation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
peroperative opioid consumption | opioid consumption during surgery
  In addition to the standard monitoring , we associate that of narcosis (BIS, Covidien LLC.Mansfield, USA) whose level is maintained between 40 and 60, a monitoring of the capnia, maintained between 35 and 40mmHg, we associate an analyzer of gas.The maintenance of the anesthesia is provided by sevoflurane adjusted according to the values of the bi-spectral index. Remifentanil is administered by the electrical pump as a function of the variation in blood pressure and heart rate, which should not exceed 20% of their baseline values during the surgical procedure.All our patients were operated by the same team.
  Ten minutes before closure, each patient receives 1 g of paracetamol (Perfalgan®) and 50 to 100 mg of tramadol depending on his weight. The remifentanil syringe pump is stopped when the skin is closed and the total dose is calculated for each patient.

SECONDARY OUTCOMES:
postoperative opioid consumption | first 24 hours after surgery
  the investigator proceed to evaluate pain at H0, H2, H4, H6, H12 and H24 postoperative hour. Each time the patient had a Visual analogic scale (VAS) greater than or equal to 40mm(from 0 to 100) a titration of 3 mg intravenous morphine every 5 minutes until VAS <40mm . Total dose of morphine required was calculated 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: ali majdoub, PHD, Principal Investigator — tunisian ministery of health
Locations (1):
- Mahdia University Hospital, Mahdia, Mahdia Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No